CLINICAL TRIAL: NCT05123482
Title: A Phase I/IIa Multi-center, Open-label Master Protocol Dose Escalation and Expansion Study of AZD8205 as Monotherapy and in Combination With Anticancer Agents in Participants With Advanced Solid Tumors (BLUESTAR)
Brief Title: A Phase I/IIa Study of AZD8205 Given Alone or Combined, in Participants With Advanced/Metastatic Solid Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6900C00001; 2022-502759-70-01 (Registry Identifier: CTIS (EU)); 2021-000736-66 (EudraCT Number)
Record Dates: First submitted 2021-10-13; First posted 2021-11-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Biliary Tract Carcinoma; Ovarian Cancer; Endometrial Cancer; Squamous Non-Small Cell Lung Cancer
Keywords: First In Human, antibody drug conjugate, cancer, solid tumour, Phase I, Phase IIa
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Neoplasms | interventions — AZD5305

STUDY DESIGN:
Intervention Model Description: The study consists a master protocol with sub studies each evaluating the safety and tolerability of AZD8205 dosed as monotherapy, or in Combination with Anticancer Agents in Participants with Advanced Solid Tumours:
  Sub Study 1 (AZD8205 monotherapy)
  * Part A Dose Escalation
  * Part B Dose Expansion
  Sub Study 2 (AZD8205 in combination with rilvegostomig)
  * Part A Dose Escalation
  * Part B Dose Expansion
  Sub Study 3 (AZD8205 in combination with saruparib with or without rilvegostomig)
  * Part A Dose Escalation
  * Part B Dose Expansion
  Sub Study 4 (AZD8205 in combination with AZD9574 with or without rilvegostomig)
  * Part A Dose Escalation
  * Part B Dose Expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sub-Study 1 AZD8205 Monotherapy (Experimental): Sub-Study 1 has two parts:
  Part A : The aim is to determine the safety, tolerability, Recommended Phase 2 Dose (RP2D), and/or the Maximum Tolerated Dose (MTD) of AZD8205.
  Part B: The aim of dose expansion is to evaluate anti-tumor activity of AZD8205 as monotherapy in select solid tumors.
  Interventions: Drug: AZD8205
- Sub Study 2: AZD8205 in combination with rilvegostomig (Experimental): Sub-Study 2 has two parts:
  Part A : Dose escalation to determine the safety, tolerability of AZD8205 + rilvegostomig Part B: Dose expansion to evaluate anti-tumor activity of AZD8205 + rilvegostomig in select solid tumors.
  Interventions: Drug: AZD8205 and AZD2936 (Rilvegostomig)
- Sub-Study 3 AZD8205 in combination with saruparib, with or without rilvegostomig (Experimental): Sub-Study 3 has two parts:
  Part A : Dose escalation to determine the safety, tolerability of AZD8205 + saruparib. Rilvegostomig may be added in a triplet combination once an AZD8205 + saruparib combination dose/schedule has been considered safe.
  Part B: Dose expansion to evaluate anti-tumor activity of AZD8205 + saruparib with or without rilvegostomig in select solid tumors.
  Interventions: Drug: AZD8205 and AZD5305 (saruparib); Drug: AZD8205 and AZD5305 (saruparib) and AZD2936 (rilvegostomig)
- Sub-Study 4: AZD8205 in combination with AZD9574 with or without rilvegostomig (AZD2936) (Experimental): Sub-Study 4 has two parts:
  Part A : Dose escalation to determine the safety, tolerability of AZD8205 + AZD9574. Rilvegostomig may be added in a triplet combination once an AZD8205 + AZD9574 combination dose/schedule has been considered safe.
  Part B: may be added in the future depending on emerging data, following a formal protocol amendment.
  Interventions: Drug: AZD8205 in combination with AZD9574; Drug: AZD8205 in combination with AZD9574 plus rilvegostomig (AZD2936)

INTERVENTIONS:
Drug: AZD8205 — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial cancers and squamous non-small cell lung cancers.
  Arms: Sub-Study 1 AZD8205 Monotherapy
Drug: AZD8205 and AZD2936 (Rilvegostomig) — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial cancers and squamous non-small cell lung cancers.
  Rilvegostomig is a bispecific antibody that specifically binds to human TIGIT and PD-1 and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Arms: Sub Study 2: AZD8205 in combination with rilvegostomig
Drug: AZD8205 and AZD5305 (saruparib) — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial and squamous non-small cell lung cancers.
  Saruparib is a PARP inhibitor that stops the PARP protein from doing its repair work in damaged cancer cells, resulting in cell death, and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Arms: Sub-Study 3 AZD8205 in combination with saruparib, with or without rilvegostomig
Drug: AZD8205 and AZD5305 (saruparib) and AZD2936 (rilvegostomig) — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial and squamous non-small cell lung cancers.
  Saruparib is a PARP inhibitor that stops the PARP protein from doing its repair work in damaged cancer cells, resulting in cell death, and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Rilvegostomig is a bispecific antibody that specifically binds to human TIGIT and PD-1 and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Arms: Sub-Study 3 AZD8205 in combination with saruparib, with or without rilvegostomig
Drug: AZD8205 in combination with AZD9574 — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial and squamous non-small cell lung cancers.
  AZD9574 is a PARP inhibitor that stops the PARP protein from doing its repair work in damaged cancer cells, resulting in cell death, and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Arms: Sub-Study 4: AZD8205 in combination with AZD9574 with or without rilvegostomig (AZD2936)
Drug: AZD8205 in combination with AZD9574 plus rilvegostomig (AZD2936) — AZD8205 is an antibody drug conjugate that has the potential to treat a wide variety of solid tumors including but not limited to breast cancer, Biliary Tract Cancer, ovarian, endometrial and squamous non-small cell lung cancers.
  AZD9574 is a PARP inhibitor that stops the PARP protein from doing its repair work in damaged cancer cells, resulting in cell death, and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Rilvegostomig is a bispecific antibody that specifically binds to human TIGIT and PD-1 and is a potential anticancer therapy in patients with advanced or metastatic solid tumors.
  Arms: Sub-Study 4: AZD8205 in combination with AZD9574 with or without rilvegostomig (AZD2936)

SUMMARY:
This research study is studying a new compound, AZD8205, as a possible treatment for advanced or metastatic solid tumours alone or in combination with anti-cancer agents

DETAILED DESCRIPTION:
This study is a Phase I/IIa Multi-center, Open-label Master Protocol Dose Escalation and Expansion Study of AZD8205 as Monotherapy and in Combination with Anticancer Agents in Participants with Advanced Solid Tumors

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years
* Relapsed/metastatic solid tumors treated with prior adequate standard of care therapy for tumor type and stage of disease or where in the opinion of the Investigator, a clinical trial is the best option for the next treatment based on response and/or tolerability to prior therapy.
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* Life expectancy ≥ 12 weeks
* Adequate bone marrow, hepatic, and renal function as defined in the protocol

Additional Inclusion Criteria For Sub-Study 1 Part A:

• Histologically or cytologically confirmed metastatic or locally advanced/recurrent breast cancer, ovarian cancer, BTC or endometrial cancer

Additional Inclusion Criteria For Sub-Study 1 Part B:

* Histologically or cytologically confirmed metastatic or locally advanced and recurrent disease for the respective cohort:

  1. Cohort B1 (Biliary Tract Cancer)
  2. Cohort B2 (Ovarian Cancer)
  3. Cohort B3 (Breast Cancer)
  4. Cohort B4 (Endometrial Cancer)
  5. Cohort B5 (Squamous Non-Small Cell Lung Cancer)

     Additional Inclusion Criteria For Sub-Study 2 Part A:
* Minimum body weight ≥ 30 kg.
* Histologically or cytologically confirmed metastatic or locally advanced/recurrent breast cancer, ovarian cancer, BTC, endometrial cancer or squamous non-small cell lung cancer.

Additional Inclusion Criteria For Sub-Study 3 Part A:

* Minimum body weight ≥ 30 kg (for participants enrolled in cohorts including rilvegostomig only).
* Histologically or cytologically confirmed metastatic or locally advanced/recurrent breast cancer, ovarian cancer, BTC, endometrial cancer or squamous non-small cell lung cancer.

Additional Inclusion Criteria For Sub-Study 4 Part A:

* Minimum body weight ≥ 30 kg (for participants enrolled in cohorts including rilvegostomig only).
* Histologically or cytologically confirmed metastatic or locally advanced/recurrent breast cancer, endometrial cancer or squamous non-small cell lung cancer.
* Participants must have progressed following at least one but no more than 3 prior lines of treatment for metastatic or relapsed disease and have no satisfactory alternative treatment option as judged by the Investigator.

Key Exclusion Criteria:

* Treatment with any of the following:

  1. Nitrosourea or mitomycin C within 6 weeks prior to the first dose of study treatment
  2. Any investigational agents or study drugs from a previous clinical study within 5 half-lives or 28 days (whichever is shorter) prior to the first dose of study treatment
  3. Any other anticancer treatment within the following time periods prior to the first dose of study intervention:

     1. Cytotoxic treatment: 21 days
     2. Non-cytotoxic drugs: 21 days or 5 half-lives (whichever is shorter)
     3. Biological products including immuno-oncology agents: 28 days
* Spinal cord compression or a history of leptomeningeal carcinomatosis.
* Brain metastases unless treated, asymptomatic, stable, and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent for at least 4 weeks prior to start of study.
* Active infection including tuberculosis and HBV, HCV or HIV
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Participants with any of the following cardiac criteria:

  1. History of arrhythmia which is symptomatic or requires treatment (NCI CTCAE v5.0 Grade 3); symptomatic or uncontrolled atrial fibrillation, or asymptomatic sustained ventricular tachycardia.
  2. Uncontrolled hypertension.
  3. Acute coronary syndrome/acute myocardial infarction, unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention, or coronary artery bypass grafting within 6 months.
  4. History of brain perfusion problems (eg, carotid stenosis) or stroke, or transient ischemic attack in the last 6 months prior to screening.
  5. Symptomatic heart failure (NYHA class ≥ 2).
  6. Prior or current cardiomyopathy.
  7. Severe valvular heart disease.
  8. Mean resting QTcF > 470 msec.
  9. Risk factors for QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age.
* Patients with history of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML (as determined by prior diagnostic investigation)

Additional Exclusion Criteria For Sub-Study 2 Part A:

* Thromboembolic event within 3 months before the first dose of study intervention - No longer applicable per amendment 7
* Experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* History of organ transplant

Additional Exclusion Criteria For Sub-Study 2 Part B

• Previous treatment with any therapy that contains a TOP1i (eg. irinotecan, topotecan, trastuzumab deruxtecan, etc.)

Additional Exclusion Criteria For Sub-Study 3 Part A:

* Concomitant use of medications or herbal supplements known to be strong cytochrome P (CYP) 3A4 inducers/inhibitors.
* Any history of persisting (> 2 weeks) severe cytopenia due to any cause
* Patients with any known predisposition to bleeding
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of saruparib.
* Previous treatment with any therapy that contains a TOP1i (eg. irinotecan, topotecan, trastuzumab deruxtecan, etc.)

Additional Exclusion Criteria For Sub-Study 4 Part A:

* Patients have received prior therapy with AZD9574 or more than 1 prior line of any other PARPi-based regimen
* Concomitant use of medications or herbal supplements known to be strong cytochrome P (CYP) 3A4 inducers/inhibitors.
* Previous treatment with rilvegostomig for the cohort treated with rilvegostomig
* Previous treatment with any therapy that contains a TOP1i (eg. irinotecan, topotecan, trastuzumab deruxtecan, etc.)
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9574

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
The number of patients with adverse events | From time of Informed consent to 30 days post last dose (approximately 1 year).
  Number of patients with adverse events by system organ class and preferred term
The number of patients with serious adverse events | From time of Informed consent to 30 days post last dose (approximately 1 year)
  Number of patients with serious adverse events by system organ class and preferred term
The number of patients with dose-limiting toxicity (DLT), as defined in the protocol. | From first dose of study treatment until the end of Cycle 1 (approximately 21 days).
  A DLT is defined as any toxicity that occurs from the first dose of study treatment up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation and which includes pre-defined haematological and non-haematological toxicities.
The number of patients with changes from baseline laboratory findings, ECGs and vital signs | From time of informed consent to 30 days post last dose (approximately 1 year)
  Description of laboratory findings and vital signs variables over time including change from baseline.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From first dose of AZD8205 to progressive disease or death in the absence of disease progression ( approx. 2 years )
  The percentage of patients with a confirmed investigator assessed complete or partial response according to response criteria in solid tumours (RECIST 1.1).
Duration of response (DoR) | From the first documented response to confirmed progressive disease or death ( approx. 2 years )
  The time from the date of first response until date of disease progression (RECIST 1.1) or death in the absence of disease progression.
Progression free Survival (PFS) | From first dose of AZD8205 to progressive disease or death in the absence of disease progression ( approx. 2 years )
  The time from first dose until RECIST 1.1 defined disease progression or cessation of study treatment.
Disease Control Rate at 12 weeks (DCR-12) | Measured from first dose until progression. For each patient, this is expected to be at 12 weeks
  Percentage of patients with confirmed CR or PR or having SD maintained for >= 11 weeks from first dose (RECIST 1.1).
Overall Survival (OS) | From first dose of AZD8205 to death ( approx. 2 years )
  The time from the date of the first dose of study treatment until death due to any cause.
Pharmacokinetics of AZD8205: Area Under the concentration-time curve (AUC) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  Area under the plasma concentration-time curve
Pharmacokinetics of AZD8205: Maximum plasma concentration of the study drug (Cmax) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  Maximum observed plasma concentration of the study drug
Pharmacokinetics of AZD8205: Time to maximum plasma concentration of the study drug (T-max) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  Time to maximum observed plasma concentration of the study drug
Pharmacokinetics of AZD8205: Clearance | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  A pharmacokinetic measurement of the volume of plasma from which the study drug is completely removed per unit time.
Pharmacokinetics of AZD8205: Terminal elimination half-life (t 1/2) | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  Terminal elimination half life.
Immunogenicity of AZD8205. | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  The number and percentage of participants who develop ADAs.
Sub Study 1: AZD8205 monotherapy Pharmacodynamics | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  To assess the intratumoral pharmacodynamic biomarkers (gamma H2AX H-scores) to AZD8205 when administered as a monotherapy.
Sub Study 2: AZD8205 in combination with rilvegostomig Pharmacodynamics | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 ( approx 2 years )
  To assess the change in intratumoral pharmacodynamic biomarkers (gamma H2AX H-scores) to AZD8205 when administered in combination with rilvegostomig.
Sub-study 2: Rilvegostomig Pharmacokinetics when in combination with AZD8205 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  To characterize the PK serum concentrations and PK parameters of rilvegostomig in combination with AZD8205.
Sub-study 2: Immunogenicity of Rilvegostomig when in combination with AZD8205 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  The number and percentage of participants who develop ADAs.
Sub-Study 3: Pharmacokinetics of saruparib in combination with AZD8205 with or without rilvegostomig | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  To characterize the PK plasma concentration and PK parameters of saruparib, including but not limited to AUC, Cmax, tmax, clearance, and half-life, as data allow, of saruparib when given in combination with AZD8205 with or without rilvegostomig.
Sub-study 3: Pharmacokinetics of rilvegostomig in combination with AZD8205 and saruparib | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  To characterize the PK serum concentrations and PK parameters (where applicable) of rilvegostomig when given in combination with AZD8205 and saruparib.
Sub-Study 3: Immunogenicity of rilvegostomig in combination with AZD8205 and saruparib | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  The number and percentage of participants who develop ADAs.
Sub-Study 4: Pharmacokinetics of AZD9574 in combination with AZD8205 with or without rilvegostomig | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  To characterize the PK plasma concentration and PK parameters of AZD9574, including but not limited to AUC, Cmax, tmax, clearance, and half-life, as data allow, of AZD9574 when given in combination with AZD8205 with or without rilvegostomig.
Sub-study 4: Pharmacokinetics of rilvegostomig in combination with AZD8205 and AZD9574 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  To characterize the PK serum concentrations and PK parameters (where applicable) of rilvegostomig when given in combination with AZD8205 and AZD9574.
Sub-Study 4: Immunogenicity of rilvegostomig in combination with AZD8205 and AZD9574 | From the first dose of study intervention, at predefined intervals throughout the administration of AZD8205 (approx 2 years)
  The number and percentage of participants who develop ADAs.

CONTACTS AND LOCATIONS:
Locations (60):
- United States (15):
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Sarasota, Florida
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Commack, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Clayton
  - Research Site, Melbourne
  - Research Site, Nedlands
  - Research Site, South Brisbane
- Belgium (2):
  - Research Site, Anderlecht
  - Research Site, Leuven
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (6):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Kunming
  - Research Site, Shandong
- Research Site, Budapest, Hungary
- Italy (4):
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (6):
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Sunto-gun
- Research Site, Amsterdam, Netherlands
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
- Taiwan (3):
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Huang Y, Tan HY, Yuan J, Mu R, Yang J, Ball K, Vijayakrishnan B, Masterson L, Kinneer K, Luheshi N, Liang M, Rosenbaum AI. Extensive Biotransformation Profiling of AZD8205, an Anti-B7-H4 Antibody-Drug Conjugate, Elucidates Pathways Underlying Its Stability In Vivo. Anal Chem. 2024 Oct 22;96(42):16525-16533. doi: 10.1021/acs.analchem.4c02309. Epub 2024 Oct 11. PMID 39392424
- See also: First in Human Study to Evaluate AZD8205 — https://www.breastcancerstudylocator.com/trial/listing/311155